CLINICAL TRIAL: NCT07037563
Title: Developing an AI Pharmacy Chatbot for the Population of Hong Kong
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Laboratory of Data Discovery for Health (Unknown); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Joseph Tsz Kei Wu, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UW 23-518
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hyperglycaemia; Hypertension; Hyperlipidaemia; Artificial Intelligence (AI)
Keywords: Chatbot; Intelligent Conversational Agent; Artificial Intelligence; Implementation Science
MeSH Terms: conditions — Hyperglycemia; Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacy chatbot intervention group (Experimental): In this arm, participants will receive a pharmacy chatbot intervention. They will be invited to use the chatbot through WhatsApp. They can ask questions regarding their (or the patient they are caring for) prescribed medications and get immediate responses from the chatbot. The intervention will last for 7 days.
  Interventions: Other: An AI pharmacy chatbot offering information related to HA-prescribed medication for hyperglycaemia, hypertension, and hyperlipidaemia
- Control group (No Intervention): The control group will not have any exposure with the chatbot during the intervention period.

INTERVENTIONS:
Other: An AI pharmacy chatbot offering information related to HA-prescribed medication for hyperglycaemia, hypertension, and hyperlipidaemia — It is a chatbot for HA-prescribed medication used for treating hyperglycaemia, hypertension, and hyperlipidaemia, available through WhatsApp. All the responses will be extracted from a database, in which the content was obtained from and validated by pharmacists from the Chief Pharmacist's Office of the Hospital Authority in Hong Kong. The intervention period will last for 7 days.
  Arms: Pharmacy chatbot intervention group

SUMMARY:
The primary objective of this study is to is to develop a conversational AI service (chatbot) in Hong Kong to assist patients and caregivers with inquires related to Hospital Authority (HA)-prescribed medications, and to evaluate its effectiveness in answering medication-related questions. The main questions it aims to answer are:

1. How satisfied are the patients and caregivers with this pharmacy chatbot?
2. How will the pharmacy chatbot impact eligible patients or caregivers on their (or the patient they are caring for) medication adherence, knowledge, and the consultation time with HA pharmacists?

There will be an intervention group and a control group:

1. The intervention group will be invited to use the AI Pharmacy Chatbot online for 7 days through WhatsApp, a commonly used social media platform in Hong Kong. They can inquire about their medications prescribed under HA and get instant, validated answers from the chatbot.
2. The control group will not use the chatbot during the intervention period.

To evaluate the chatbot's usability, researchers will measure patient satisfaction through usability questionnaires issued to the intervention group after their intervention period. Differences in medication adherence, medication knowledge, and HA pharmacist consultation time will also be measured between the intervention and control groups after the intervention period, to determine the chatbot's impact.

DETAILED DESCRIPTION:
In this study, we aim to develop an artificial intelligent (AI) pharmacy chatbot and evaluate its effectiveness in answering questions related to prescribed-medications.

We will first develop an AI pharmacy chatbot prototype utilizing advanced technologies such as AI and natural language processing. By implementing Hospital Authority (HA) drug database and suggestions from Chief Pharmacist's Office (CPO), a Proof-of-Concept phase will be conducted to validate the chatbot's ability to address medication-related questions for locally prevalent chronic conditions in Hong Kong: hyperglycaemia, hypertension, and hyperlipidaemia. After completing the prototype development, we will invite pharmacists from HA for testing and evaluation of the prototype, further finetuning the chatbot based on their feedback.

Then we aim to enhance the usability of the chatbot by incorporating feedback from patients and caregivers. We aim to recruit a minimum of 280 patients receiving HA-prescribed medication on hyperglycaemia, hypertension, and / or hyperlipidaemia, or their caregivers. According to a previous study, the medication adherence of patients with chronic conditions in Hong Kong was about 61.63%. For an increase to 80% of adherence would require a minimum of 140 participants per group, with a significance level (α) of 0.05, a test power (1-β) of 0.8, and a cluster design effect (D) of 1.5.

Recruitment of patients and caregivers will involve collaboration with HA to identify eligible participants. Designated pharmacists and other healthcare professionals from HA will help distribute recruitment materials to eligible patients and caregivers and provide researchers a list of participants who express the willingness to participate.

Participants will be randomized in a 1:1 ratio to either the control group or the intervention group. Before the intervention period, they will all receive a consent form and an information sheet which provides details on the study. They will also be asked to complete a pre-study survey, which includes questions on socio-demographics, drug usage habits, medical history and experience with chatbots.

Participants in the intervention group will then be invited to use the pharmacy chatbot and receive a usability test guideline, with an emphasis on the chatbot's role as a support tool for medication inquiries. The intervention duration will last for 7 days and the control group will have no exposure to the chatbot during the period. After 7 days, a post-study survey will be conducted to all participants in both the intervention and control groups. Participants in the intervention group will also receive a usability questionnaire to feedback on the chatbot.

A convergent mixed methods design, combining qualitative and quantitative approaches, will be used to evaluate the intervention effect of the chatbot.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older diagnosed with either hyperglycaemia, hypertension, or hyperlipidaemia, and currently receiving medication prescribed by the Hospital Authority in Hong Kong.
* Caregivers aged 18 years or older for patients described above.

Exclusion Criteria:

* There is no exclusion criterion, but they should meet the inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Medical knowledge | 1 week
  Before the intervention period, all participants will be asked whether they disagree or agree with the following statements on a 5-point Likert scale (Strongly agree, Agree, Neutral, Disagree and Strongly disagree):
  1. I understand the main indications of my medications (or the medications of the patient I care for).
  2. I understand the potential side effects of my medications (or the medications of the patient I care for).
  3. I know how to take my medications (or administer the medications of the patient I care), including the dosage and frequency, thereby promoting my medication adherence.
  4. I have concerns or worries about my medications (or the medications of the patient I care for).
  5. I can obtain medication-related information efficiently and easily.
  After the 7-day intervention period, they will be asked again the same questions.
Medical adherence | 1 week
  Before the intervention period, all participants will be asked whether they disagree or agree with the following statement on a 5-point Likert scale (Strongly agree, Agree, Neutral, Disagree and Strongly disagree): I know how to take my medications (or administer the medications of the patient I care), including the dosage and frequency, thereby promoting my medication adherence.
  After the 7-day intervention period, they will be asked again the same questions.

SECONDARY OUTCOMES:
Response time | 1 week
  We will calculate from the backend the chatbot's response time when responding to user's input (text, image and voice).
User satisfaction | 1 week
  Participants in the intervention group will be asked whether they disagree or agree to the following statements on a 5-point Likert scale (Strongly disagree, Disagree, Neutral, Agree and Strongly agree):
  1. The chatbot is simple to use and user-friendly.
  2. The chatbot understands my queries and is able to address them.
  3. The chatbot's responses are relevant and sufficient.
  Moreover, they will also be asked to rate their overall experience with the chatbot on a 5-point Likert scale (Very Good, Good, Moderate, Poor, and Very Poor), and whether they will use the chatbot again in the future and whether they would recommend others to use the chatbot.
Consultation with pharmacists | 1 week
  Before the intervention period, we will ask all participants their frequency and consultation time with pharmacists. After the 7-days intervention period, we will ask them again whether they have visited any pharmacists during the time, and if so, the frequency and consultation time.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Wu, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Laboratory of Data Discovery for Health, Hong Kong
  - The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after de-identification (text, tables, figures, and appendices), will be shared. A written data-sharing request for meta-analysis should be submitted by email with a methodologically sound proposal. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal for meta-analysis. To gain access, data requestors will need to sign a data access agreement.